CLINICAL TRIAL: NCT04753918
Title: Single Center, Prospective, Open Label, Single-arm Clinical Study of Safety & Feasibility of Using Navigational Bronchoscopy to Perform Interstitial PD Therapy Using Lipiodol® as a Light Deliver and Photofrin® as Treatment in Subjects With Unresectable Solid Tumor in Peripheral Lung
Brief Title: Novel Light Delivery Methods for Lung Cancer Photodynamic Therapy - A Pilot Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYGH107071
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Lung Metastasis
Keywords: Photodynamic Therapy; Peripheral Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dihematoporphyrin Ether; Ethiodized Oil; Optical Fibers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Novel light delivery methods for photodynamic therapy (Experimental): High refraction-index contrast medium: Lipiodol injected in the bronchial tree can enhance the treatment extension of the photodynamic therapy
  Interventions: Drug: Porfimer sodium; Drug: Ethiodized oil; Procedure: Novel light delivery methods of photodynamic therapy; Device: Fiber optic

INTERVENTIONS:
Drug: Porfimer sodium — Photofrin 2mg/kg was iv injected 48-50 hours before light illumination.
  Other Names: Photofrin
Drug: Ethiodized oil — In hybrid operation room setting, a navigational bronchoscope guide sheath was inserted to the proximal end of the tumor region. About 5 ml Lipiodol was infused to full cover whole the tumor.
  Other Names: Lipiodol
Procedure: Novel light delivery methods of photodynamic therapy — Using high-refraction index contrast medium: lipiodol as a light diffusor to enhance the range of photodynamic therapy
Device: Fiber optic — A cylindrical laser fiber was then inserted through the guide sheath to the tumor region then illuminate light to complete the photodynamic therapy.

SUMMARY:
This research study is being conducted to assess the safety and feasibility of using a newly developed bronchoscopic light delivery method of photodynamic therapy to treat subjects with solid tumors in peripheral lung, who are inoperable or refused surgery.

DETAILED DESCRIPTION:
Lung cancer accounts for almost one-third of cancer deaths. Cancer screening strategies have the potential to achieve a 20% reduction in death rates. Newly developed bronchoscopic technologies (such as navigational bronchoscopy in a hybrid operation room) have been shown to enable physicians to safely reach lesions in peripheral regions of the lung and obtain a diagnosis. This new technology may now potentially offer bronchoscopic therapeutic interventions, such as photodynamic therapy, to tumors that were previously unreachable due to their peripheral anatomic location.

Photodynamic therapy (PDT) uses a combination of a photosensitizing drug (a drug that is activated by light), called porfimer sodium (Photofrin®), and a light from a laser that emits no heat. This technique works to allow the medical doctor to specifically target and destroy abnormal or cancer cells while limiting damage to surrounding healthy tissue. The activation of the drug is done by lighting the abnormal area using a fiber-optic device (very fine fiber [like a fishing line] that permits light transmission) inserted into a flexible tube called a bronchoscope. The light activates the porfimer sodium, which is concentrated in the abnormal tissue, leading to its destruction. But the penetrating depth of light is about 1.5 to 2 cm limits the treatment range of tumor size.

We proposed a novel light delivery method of instilling a high-refractive-index (RI) liquid (Lipiodol) to enhance light delivery in the lung.

The purpose of this study is to determine if physicians can reach the tumors in the periphery of the lung via electro-navigational bronchoscopy in a hybrid operation room and inject the lipiodol to cover the whole tumor then deliver photodynamic therapy by placing the optical fiber into the tumor

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 20 and 75
* Diagnosed with histologically confirmed solid tumor located in the peripheral lung
* Not candidate or failed of standard chemotherapy, radiotherapy or surgery
* Primary lung cancer without mediastinal or distant lymph nodes metastasis (N0-N1)
* The tumor is ≤ 2 cm in size and clearly observable in computerized tomography (CT scan)
* Able to sign an informed consent

Exclusion Criteria:

* Diagnostic of small cell lung cancer or non-solid malignancy
* Solid tumor located in central lung
* Primary lung cancer without distant metastasis (M0)
* Received radiotherapy over the target tumor
* Abnormal blood results
* Received chemotherapy/immunotherapy in the last 4 weeks
* Tumor invasion with major blood vessels
* Allergy to porphyria or known hypersensitivity to Photofrin® or porphyrin-like compounds or to any of its excipients, allergy to Lipiodol or iodine-content contrast medium
* Planned surgical procedure within the next 90 days
* Coexisting ophthalmic disease likely to require slit-lamp examination within the next 90 days
* Acute or chronic medical or psychological illnesses that prevent endoscopy procedures
* Pregnant or intend to become pregnant, breastfeeding or intend to breastfeed during the study
* Received PDT during the past 1 months
* Severe impairment of your kidney or liver function
* Participates or intends to participate in another drug study (other than observational studies) during the study
* Victim of AIDS
* Other critical condition that the investigator considered not suited for participation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility to Perform Novel Photodynamic Therapy Into Tumor | Day 3 post-treatment
  Number of times photodynamic therapy was delivered into the tumor using navigational bronchoscopy for each subject.
Adverse Events Incidence Indicating Safety of Novel Photodynamic Therapy | Up to 6 months
  The incidence of adverse events following Novel PDT will be presented as the primary safety indicator for this treatment.

SECONDARY OUTCOMES:
Tumor Response at 3 Months Post Photodynamic Therapy (PDT) | Up to 3 months
  From the start of treatment until 3 months post-treatment measured as per the Modified RECIST (Response Evaluation Criteria in Solid Tumors) Criteria
Tumor Response at Study Exit (6 Months) Post Photodynamic Therapy (PDT) | From the start of treatment until 6 months post-treatment measured as per the Modified RECIST (Response Evaluation Criteria in Solid Tumors) Criteria
  Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yei-San Hsieh, MD, Principal Investigator — Taoyan General Hospital, Ministry of Health and Welfare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang H, Liao KS, Hsieh YS. Bronchoscopic light delivery method for peripheral lung cancer photodynamic therapy. J Thorac Dis. 2020 Jul;12(7):3611-3621. doi: 10.21037/jtd-19-3887. PMID 32802440
- [Result] Friedberg JS, Skema C, Burdick J, Yodh AG, Carr SR, Culver JP. A novel technique for light delivery through branched or bent anatomic structures. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1963-7. doi: 10.1016/s0022-5223(03)01320-5. PMID 14688713
- [Result] Chen KC, Lee JM. Photodynamic therapeutic ablation for peripheral pulmonary malignancy via electromagnetic navigation bronchoscopy localization in a hybrid operating room (OR): a pioneering study. J Thorac Dis. 2018 Apr;10(Suppl 6):S725-S730. doi: 10.21037/jtd.2018.03.139. PMID 29732193
- See also: Feasibility Study of Using Navigational Bronchoscopy to Perform PDT-Photofrin® in Unresectable Peripheral Lung Cancer — https://clinicaltrials.gov/ct2/show/results/NCT02916745